CLINICAL TRIAL: NCT05265936
Title: Is it Safe to Advance a Guidewire Through a Previously Deployed Double j Stent? A Prospective, Randomized, Controlled Study
Brief Title: Is it Safe to Advance a Guidewire Through a Previously Placed Double j Stent?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DJG2022
Record Dates: First submitted 2022-02-22; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Kidney Stone; Ureter Obstruction; Stent Complication
Keywords: double j stent; guidewire; infection
MeSH Terms: conditions — Kidney Calculi; Ureteral Obstruction; Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidewire through DJ stent (Active Comparator): Patients who underwent lithotripsy after guidewire insertion through a previously placed double j stent.
  Interventions: Procedure: Passing a guidewire through a double j stent
- DJ stent remove + guidewire (Sham Comparator): Patients who underwent lithotripsy after double j stent removal and guidewire placement.
  Interventions: Procedure: Double J stent removal and guidewire insertion

INTERVENTIONS:
Procedure: Passing a guidewire through a double j stent — The previously placed double J stent is removed up to the urethral meatus with a cystoscope and forceps and kept fixed at the meatal level without further pulling. Then, after reaching the kidney by passing a guidewire through it, the double j stent is removed. Followed by the routine lithotripsy procedure.
  Arms: Guidewire through DJ stent
Procedure: Double J stent removal and guidewire insertion — The double j stent is completely removed with the cystoscope and forceps, and the guidwire is inserted into the ureter by visualizing it with the cystoscope. Followed by the routine lithotripsy procedure.
  Arms: DJ stent remove + guidewire

SUMMARY:
In this prospective randomized controlled study, it is aimed to investigate the effects of guidewire advanced through a previously placed double j stent on postoperative complications, operation time and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Double J stent placed at least 2 weeks ago

Exclusion Criteria:

* Active urinary tract infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complication | 3 months
  Rate of patients who had a postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

REFERENCES:
- [Background] Leslie SW, Sajjad H. Double J Placement Methods Comparative Analysis. 2023 May 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482453/ PMID 29494060